CLINICAL TRIAL: NCT05705726
Title: Ultrasound Guided Fascia Iliaca Block Versus Intravenous Dexmedetomidine and Ketamine for Positioning Fracture Femur Patients During Spinal Anesthesia: Randomized Comparison Study
Brief Title: Fascia Iliaca Block Versus Intravenous Dexmedetomidine and Ketamine for Positioning Fracture Femur
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 524/2022
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Pain; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Infusion Pumps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- facia iliaca block (Experimental)
  Interventions: Device: ultrasound guided facia iliaca block
- Precedex and ketamine (Experimental)
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Device: ultrasound guided facia iliaca block — Patient will received ultrasound guided fascia iliaca block by 20 ml Bupivacaine 0,25% .
  Arms: facia iliaca block
Drug: Intravenous drug — Patient will received intravenous injection of precedex 0.25mic/Kg and ketamine 0,2 mg/kg .
  Arms: Precedex and ketamine

SUMMARY:
Proximal femur fractures are one of the commonest fractures especially in the elderly population. Early surgical fixation is the best analgesic for associated pain. Spinal anesthesia has been favored by many anesthesiologists due to the simplicity of the technique, the better analgesic profile, and the lower incidence of complications like delirium and thromboembolic events. However, severe pain, encountered during positioning for spinal anesthesia, can complicate the technique and worsen the patient experience.

the study aim to compare the analgesic effect of intravenous dexmedetomidine and fascia iliaca block preoperatively to assist positioning patients for performance of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years.
2. Hip fractures
3. Both sexes.

Exclusion Criteria:

1. Patient refusal
2. Allergy to local anesthetics
3. Bleeding diathesis or history of anticoagulant use.
4. impaired cognition or dementia
5. . Infection of the skin at the site of needle punctures area
6. multiple fractures
7. Any previous analgesic administration during the last 12 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral pain scale | during spinal anesthesia
  0 = calm, 1 = facial grimacing, 2 = moaning, 3 = screaming, and 4 = unable to proceed because of restlessness or agitation

SECONDARY OUTCOMES:
Quality of patient's position | before spinal anesthesia
  0 = poor hip flexion, 1 = satisfactory hip flexion, 2 = good hip flexion, and 3 = optimal hip flexion

CONTACTS AND LOCATIONS:
Overall Officials: hassan m. hetta, lecturer, Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No